CLINICAL TRIAL: NCT03242473
Title: Mitigating the Inflammatory Response in Acute Pancreatitis With Appropriate Fluid Management; A Randomized Clinical Control Trial Comparing the Effects of Lactated Ringers and Normal Saline
Brief Title: Comparing the Effects of Lactated Ringers and Normal Saline in Acute Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Children's National Research Institute (Other); Children's Hospital of The King's Daughters (Other)
Responsible Party: Principal Investigator, Peter Farrell, Clinical Fellow, Department of Pediatrics, Division of Gastroenterology, Hepatology and Nutrition, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-12-FB-0245
Record Dates: First submitted 2016-08-22; First posted 2017-08-08 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactated Ringers (LR) (Experimental): The subject will be placed on 1.5x maintenance IVF with the fluids to which they are randomized. Fluid Management will be the intervention.
  Interventions: Other: Fluid Management
- Normal Saline (NS) (Experimental): The subject will be placed on 1.5x maintenance IVF with the fluids to which they are randomized. Fluid Management will be the intervention.
  Interventions: Other: Fluid Management

INTERVENTIONS:
Other: Fluid Management — The patient will remain NPO for at least the first 24 hours. The following studies will be obtained at the time of admission if not previously obtained in the ED: CMP, GGT, Amylase, Lipase, Triglycerides, CBC, and CRP, along with an abdominal ultrasound. CBC, CRP, BMP, amylase and lipase levels will be obtained at 24 and 48 hours (+/- 2 hours). SIRS status will be evaluated with vital sign checks every 4 hours and the leukocyte counts every 24 hours.
  Other Names: Resuscitative fluids for acute pancreatitis

SUMMARY:
Acute pancreatitis is increasingly common diagnosis in children. Most of the guidelines related to the details of management of acute pancreatitis are extrapolated from the adult literature. There is only limited data regarding management of acute pancreatitis in children. The mainstay of management is bowel and pancreatic rest with significant fluid support to minimize the effect of the cytokines on the pancreas and other organs. The standard fluid choices are Lactated Ringer's solution (LR) and normal saline (NS). Currently, both LR and NS are used at the discretion of the treating physician as the standard of care for acute pancreatitis. The investigators hope to examine the question of ideal fluid choice for fluid resuscitation in children with acute pancreatitis by assessing recovery time in the context of measured inflammatory markers and SIRS status at 24 and 48 hours after admission. The ideal fluid choice in the initial resuscitation of acute pancreatitis has not been effectively evaluated before in the pediatric population. Even if there is no statistically significant difference between the two fluid options, this trial will still provide clinically significant information.

DETAILED DESCRIPTION:
Acute pancreatitis represents inflammation of the pancreas that has been well identified in the literature for several centuries. However, the phenomenon has only relatively recently gained prominence in the pediatric literature. The incidence can be as high as 13 per 100,000 per year, a level which approaches that seen in adults, and the diagnosis has been increasingly common over the last two decades. It affects all ages of children (including infants) evidenced by well-established age appropriate diagnostic criteria. The precise pathophysiological basis of the inflammation is not always as clear. Currently, the prevailing theory is that there is an insult to the acinar cells of the pancreas likely via an atypical calcium signal that releases a cascade of cellular activity and that ultimately results in a disseminated cytokine storm. While there is certainly debate as to the inciting event to this cascade, one thing that is clear is that extensive end-organ damage can occur if this cytokine storm reaches systemic circulation. Therefore, the mainstay of management is bowel (and specifically pancreatic) rest with significant fluid support to minimize or mitigate the effect of the cytokines on the pancreas and other systemic organs such as the lungs, heart, and kidneys. The remainder of therapy consists of appropriate analgesia and antiemetics.

Unfortunately, most of the guidelines related to the details of management of acute pancreatitis are extrapolated from the adult literature. There is only limited data regarding management of acute pancreatitis in children. Recently, Wu et al. have shown compelling data that suggest the choice of fluid for management of acute pancreatitis in adults should be Lactated Ringers (LR). Their group demonstrated in a small randomized controlled trial involving 40 adult patients with acute pancreatitis, that the patients randomized to the LR arm of the study had significantly lower levels of C-reactive protein and Systemic Inflammatory Response Syndrome (SIRS) markers compared with controls in the normal saline (NS) group. They proposed that the mechanism for this difference may be related to the more balanced pH of LR which might prevent, or at least further buffer, the systemic inflammation that is triggered by the release of the offending cytokines from the pancreas. Currently, both LR and NS are used at both Children's Hospital of The King's Daughters (CHKD) and Children's National Health System (CNHS) at the discretion of the attending physician as the standard of care for acute pancreatitis. The investigators hope to examine the question of ideal fluid choice for fluid resuscitation in children with acute pancreatitis by assessing recovery time in the context of measured inflammatory markers and SIRS status at 24 and 48 hours after admission.

This is a prospective randomized trial of pediatric patients in the emergency department (ED) or inpatient ward diagnosed with acute pancreatitis. Patients meeting the study inclusion criteria will be identified by an ED or inpatient physician. The ED or inpatient physician will ask the eligible patient/parent if they are interested in hearing about the study. If the eligible patient/parent is interested in hearing information about the study, the ED or inpatient ward will notify the PI via telephone or page. The PI will come to the eligible patient's room to explain the study and answer any questions, or the PI will page a research team member to do so. If the patient/parent agrees to participate in the study, the research team member will consent the parents of the patients aged 0-17 years or consent patients aged 18 years. Assent will be obtained from patients aged 8-17 years. Non-English speaking patients/parents will be consented using an in-person translator or the blue phone translating service. These consent and assent forms will be signed by a witness. At the time of enrollment, the subject identification (ID) number and medical record number will be entered into the electronic Subject ID Key. Once the patient is enrolled in the study, their treatment will be randomized to either the LR or the NS group. Both treatments are current standard of care for acute pancreatitis. Patients who choose not to participate in the study will receive the standard of care treatment at the discretion of the attending physician, which may involve either fluid, and will likely include most (if not all) of the lab studies as outlined in this protocol.

The goal is to screen and enroll the subjects in either the ED or inpatient ward within 6 hours of diagnosis, as this is within the theoretical window prior to the development of systemic inflammation. At the discretion of the attending physician, however, treatment can begin in the ED or inpatient ward before enrollment in the study; patients will not have to wait for necessary treatments. Patients will still be eligible to participate in the study if treatment was begun in the ED or inpatient ward. The randomized treatment may end up being the same or different than what was originally ordered by the attending physician. If any such changes in treatment plan are noted, this will be considered for the data analysis.

The randomization plan will include constrained randomization using the permuted blocks method. The research team member will open the envelope that contains the randomized treatment and the Admission Order Sheet that details the orders that need to be placed on admission. The research team member will communicate this information to the ED or inpatient attending physician or staff member overseeing the patient's care at the time of enrollment. All clinical treatments described in this protocol, including labs orders, are the current standard of care for acute pancreatitis diagnosis. The purpose of the Admission Order Sheet is to standardize the timeline of the lab work at admission, at 24 hours and 48 hours after admission, not to request any additional lab work for the purposes of the study.

The subject will be placed on 1.5x maintenance IVF with the fluids to which they are randomized. The patient will remain nil per os (NPO) for at least the first 24 hours, and the time of initiating feeds after 24 hours will be at the discretion of the admitting team. As the standard of care, the following studies will be obtained at the time of admission if not previously obtained in the ED: Complete Metabolic Panel (CMP), gamma-glutamyltransferase (GGT), Amylase, Lipase, Triglycerides, Complete Blood Count (CBC), and CRP, along with an abdominal ultrasound. CBC, CRP, amylase and lipase levels will be obtained at 24 and 48 hours (+/- 2 hours) as listed in the Admission Order Sheet. Similarly, a Basic Metabolic Panel (BMP) will be collected at 24 and 48 hours (+/- 2 hours), with the addition of liver function tests if liver enzyme levels are elevated at admission (as defined by transaminases greater than 2 times the age appropriate upper limit of normal). SIRS status will be evaluated with vital sign checks every 4 hours and the leukocyte counts every 24 hours.

The patients will be observed for additional known signs and complications of acute pancreatitis such as persistent inflammation, shock, sepsis, electrolyte abnormalities, renal failure or other end organ damage. Any adverse reactions during the trial will be treated independent of the trial, and the attending physician will continue to manage the care of the patient at their discretion. Any serious adverse reactions will be documented clinically and reported to the CHKD or CNHS incident reporter systems, Eastern Virginia Medical School (EVMS) Institutional Review Board (IRB), CNHS IRB and CHKD Human Research Coordination (HRC) Committee .

The de-identified information will be collected from the patient's electronic medical record by a research team member and entered directly into an Excel database. Patients transferred from an outside ED should already have charts scanned into the Electronic Health Record (EHR) as standard of care. If only a paper chart is available for any transferred patient, a research team member will enter information directly from the paper chart into the Excel database.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0-18 years diagnosed with acute pancreatitis in the emergency department or inpatient ward at Children's Hospital of The King's Daughters or one of the affiliated institutions participating in the study.

Exclusion Criteria:

* Patients greater than 18 years of age
* Patients who are not diagnosed with acute pancreatitis
* Patients who have any previous history of acute pancreatitis, past medical history of underlying illness including congenital heart disease, chronic lung disease, or renal failure
* Patients who have any of the following: hyperkalemia, systemic acidosis, acute dehydration, extensive tissue breakdown, adrenal insufficiency, concomitant use of potassium-sparing diuretics, use of extended-release preparations in patients with esophageal compression caused by an enlarged left atrium, hypersensitivity to sodium chloride, hypernatremia, or fluid retention
* Patients who are pregnant females
* Patients who have additional comorbidities at time of admission that would prevent adequate treatment with the methods described above will be excluded

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2014-12; Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
C-Reactive Protein (CRP) | At admission, 24 and 48 hours
  Primary marker of inflammation, change measured at baseline and then every 24 hours for 48 hours

SECONDARY OUTCOMES:
Blood Urea Nitrogen (BUN) | At admission, 24 and 48 hours
  Trend BUN
Serum Amylase | At admission, 24 and 48 hours
  Trend Amylase over the course of the admission
Serum Lipase | At admission, 24 and 48 hours
  Trend Lipase over the course of the admission
Average length of stay | Total length of stay in the hospital, measured in hours, usually around 4 days (96 hours).
  Total length of stay in the hospital
Time to initiation of enteral feeds | Total length of time to initiate feeds in the hospital, measured in hours, usually around 2 days (48 hours).
  Total time required to start oral feeds as defined by placement of order to start feeds
SIRS Criteria | At admission, 24 and 48 hours
  Signs of Systemic Inflammatory Response Syndrome (SIRS) as defined by Goldstein et al will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Farrell, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Sona Sehgal, MD, Principal Investigator — Children's National Research Institute; Rana Ammoury, MD, Principal Investigator — Children's Hospital of The King's Daughters; Maisam Abu-El-Haija, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - Children's National Health System, Washington D.C., District of Columbia
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of The King's Daughters, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the de-identified data obtained at CCHMC with our partners at CHKD and Children's National Medical Center, and we intend to have them share their data with us as well.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be shared for up to 3 years after the conclusion of recruitment.

REFERENCES:
- [Background] Srinath AI, Lowe ME. Pediatric pancreatitis. Pediatr Rev. 2013 Feb;34(2):79-90. doi: 10.1542/pir.34-2-79. No abstract available. PMID 23378615
- [Background] Sarr MG. Early fluid "resuscitation/therapy" in acute pancreatitis: which fluid? What rate? What parameters to gauge effectiveness? Ann Surg. 2013 Feb;257(2):189-90. doi: 10.1097/SLA.0b013e318280e19e. No abstract available. PMID 23291660
- [Background] Meyer A, Coffey MJ, Oliver MR, Ooi CY. Contrasts and comparisons between childhood and adult onset acute pancreatitis. Pancreatology. 2013 Jul-Aug;13(4):429-35. doi: 10.1016/j.pan.2013.06.005. Epub 2013 Jun 27. PMID 23890143
- [Background] Wu BU, Hwang JQ, Gardner TH, Repas K, Delee R, Yu S, Smith B, Banks PA, Conwell DL. Lactated Ringer's solution reduces systemic inflammation compared with saline in patients with acute pancreatitis. Clin Gastroenterol Hepatol. 2011 Aug;9(8):710-717.e1. doi: 10.1016/j.cgh.2011.04.026. Epub 2011 May 12. PMID 21645639
- [Background] Goldstein B, Giroir B, Randolph A; International Consensus Conference on Pediatric Sepsis. International pediatric sepsis consensus conference: definitions for sepsis and organ dysfunction in pediatrics. Pediatr Crit Care Med. 2005 Jan;6(1):2-8. doi: 10.1097/01.PCC.0000149131.72248.E6. PMID 15636651
- [Derived] Farrell PR, DesPain AW, Farmer P, Farrell LM, Greenfield B, Rogers ME, Hornung L, Kim E, Pearman R, Neway B, Thompson T, Heubi JE, Sehgal S, Amoury R, Abu-El-Haija M. Faster discharge with lactated ringers than normal saline in first 72 h of acute pancreatitis: A multicenter randomized trial. J Pediatr Gastroenterol Nutr. 2024 Feb;78(2):360-368. doi: 10.1002/jpn3.12082. Epub 2023 Dec 11. PMID 38374568